CLINICAL TRIAL: NCT01524445
Title: Retrospective Evaluation of Re-Treatment With Bortezomib in Subjects With First Relapse After Bortezomib First-Line Therapy
Brief Title: Retrospective Survey of Re-treatment With Bortezomib
Status: Completed | Type: Observational
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: EMEA Medical Affairs Director Oncology, Janssen-Cilag G.m.b.H, Germany
Other Study IDs: CR018175; 26866138MMY4053 (Other: Janssen CTMS ID)
Record Dates: First submitted 2011-06-16; First posted 2012-02-02 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Hematological Cancer; Multiple Myeloma
Keywords: Bortezomib; Velcade; multiple myeloma; retrospective study, response rate, medical resource utilization
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- bortezomib retreatment: bortezomib retreatment due to relapse Patients who received bortezomib-containing chemotherapy as first-line treatment for MM experienced partial response or better and were re-treated (second-line) with bortezomib (for at least 3 cycles) due to a relapse of the disease after a treatment free interruption of at least 6 months
  Interventions: Other: bortezomib retreatment due to relapse

INTERVENTIONS:
Other: bortezomib retreatment due to relapse — Patients who received bortezomib-containing chemotherapy as first-line treatment for MM, experienced partial response or better, and were re-treated (second-line) with bortezomib (for at least 3 cycles) due to a relapse of the disease after a treatment free interruption of at least 6 months

SUMMARY:
The purpose of this retrospective study is to collect information about patients who received bortezomib as their first chemotherapy and who responded well to it, but who relapsed afterwards and were treated again with bortezomib a second time after a treatment-free period of at least 6 months. During this non-interventional study (this means that no drug is being tested in this study) the safety and effectiveness (whether it works or not) of bortezomib re-treatment will be evaluated in patients with multiple myeloma. Only data already mentioned in your clinical file will be collected. About 100 adult patients will take part in the study

DETAILED DESCRIPTION:
This is an international, multicenter, non-interventional, retrospective study to evaluate the efficacy and safety of bortezomib in 100 adult patients diagnosed with multiple myeloma (MM) who responded to bortezomib as first-line treatment, experienced partial response or better, presented with relapsed disease, and were re-treated (second-line) with bortezomib (for at least 3 cycles) after a treatment-free interruption of at least 6 months. As this is a non-interventional study, no changes to the current treatment that the patient receives will be required, and no additional treatment will be provided by the company. The decision of the patients to take part in this study will not have any impact on the care they receive. All the appropriate treatment-related decisions will have been made by the treating physician(s), and only data available from clinical practice will be collected. Retrospective data will be collected at a single time point for each patient (the data collection visit). Each investigator should collect data from patients fulfilling all inclusion and exclusion criteria. After receiving the signed informed consent form (ICF) from the patient (if required by local regulations), the investigator will start documenting the retrospective data for each patient using electronic data capture (eDC). After confirmation of the patient's eligibility, the patient's last visit, patient characteristics, predefined risk factors (if available), MM-related data, and first- and second-line bortezomib-related data will be documented in the Case Report Form (CRF). The patient's status after re-treatment with bortezomib, medical resource utilization data, as well as (serious) adverse drug reactions ([S]ADRs) will be collected. No blood, urine, or other biological samples will be taken, and no additional investigations will be performed. the current therapy of the patient will be maintained with no changes

ELIGIBILITY:
Inclusion Criteria:

* Has a current diagnosis/was diagnosed with MM or secretory MM
* Was previously treated with bortezomib-containing chemotherapy
* Responded to bortezomib as first-line treatment
* Has been re-treated with bortezomib (at least 3 cycles) due to relapse of the disease (following the first bortezomib treatment), after a treatment-free interruption of at least 6 months
* Completed bortezomib re-treatment at least 2 months ago Exclusion Criteria:
* Was a pregnant or breastfeeding woman while receiving either first-line or second-line treatment with Velcade

Has received bortezomib-containing chemotherapy for the first time following a first relapse or later

* Has participated in a clinical trial in which bortezomib was used as second-line treatment following a relapse after response to Velcade as first-line chemotherapy, and the study data are not publicly available at the time of inclusion in the current study
* Has received bortezomib as first-line therapy and was re-treated with bortezomib after first relapse in the VISTA clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinic; Hospital
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-03; Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
overall response after retreatment | Day 1
  overall response after retreatment will be assessed from initial diagnosis to the time of data collection

SECONDARY OUTCOMES:
number of medical care encounters | Day 1
  number of medical care encounters are collected retrospectively from initial diagnosis to the time of data collection
duration of medical care encounters | Day 1
  duration of medical care encounters are collected retrospectively from initial diagnosis to the time of data collection
duration of hospitalization | Day 1
  duration of hospitalizations are collected retrospectively from initial diagnosis to the time of data collection
number and character of diagnostic and therapeutic tests and procedures | Day 1
  number and character of diagnostic and therapeutic tests and procedures are collected retrospectively from initial diagnosis to the time of data collection
outpatient medical encounters and treatments | Day 1
  outpatient medical encounters and treatments are collected retrospectively from initial diagnosis to the time of data collection
safety and tolerability | Day 1
  safety and tolerability will be evaluated based on the collection of serious and non serious adverse drug reactions from initial diagnosis to the time of data collection

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.
Locations (4):
- Greece (4):
  - Alexandroupoli
  - Athens
  - Athens Attica
  - Pátrai